CLINICAL TRIAL: NCT05015803
Title: A Non-pharmacological Multi-modal Therapy to Improve Sleep and Cognition and Reduce Mild Cognitive Impairment Risk
Brief Title: Enhanced CBTi for Older Adult Sleep and Cognition
Acronym: R44
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: University of Arizona (Other); Proactive Life Inc (Industry)
Responsible Party: Principal Investigator, Orfeu M. Buxton, Elizabeth Fenton Susman Professor of Biobehavioral Health, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R44AG056250 (NIH)
Record Dates: First submitted 2021-07-16; First posted 2021-08-20 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Insomnia; Alzheimers Disease Related Dementias
Keywords: cognitive-behavioral therapy (CBT); sleep; ADRD; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: CBTi with Application, Standard TeleHealth CBTi, and Sleep Hygiene Education study groups run in parallel after randomization.
Who Masked: Participant
Masking Description: This is a single-blind study design. The therapeutic care for insomnia is synonymous with the study intervention, therefore blinding of the CBT care provider is impossible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBTi with Application (Experimental): Device-based intervention facilitation and clinician interfacing for Cognitive Behavioral Therapy for Insomnia (CBTi).
  Interventions: Combination Product: CBTi with Application
- CBTi (Active Comparator): Standard CBTi delivered via video conferencing [Zoom Health].
  Interventions: Behavioral: CBTi
- Sleep Hygiene (Active Comparator): Treatment as usual: Sleep hygiene education and training.
  Interventions: Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Combination Product: CBTi with Application — Participants randomized to this study arm will experience an attempted enhancement of standard video conferencing CBTi, that is facilitated with electronic device-based data and resources to the clinician. Noninvasive ambulatory worn and nearable devices deliver feedback of data to the clinician on an application interface. This information will be used to inform the therapeutic approach and to facilitate a living-space environment that is conducive to effective therapy.
  Other Names: Cognitive-Behavioral Therapy for Insomnia - Enhanced
  Arms: CBTi with Application
Behavioral: CBTi — Participants randomized to this study arm will experience standard CBTi that is delivered via video conferencing by a clinician, with some application interface use.
  Other Names: Cognitive-Behavioral Therapy for Insomnia - Standard
  Arms: CBTi
Behavioral: Sleep Hygiene Education — Participants randomized to this study arm will experience sleep hygiene education and training, with some application interface use.
  Arms: Sleep Hygiene

SUMMARY:
This randomized clinical trial on 60+ aged and independent-living healthy individuals with symptoms of insomnia will attempt to improve sleep and health outcomes related to sleep with enhancement of a clinical intervention, Cognitive Behavioral Therapy for Insomnia (CBTi).

DETAILED DESCRIPTION:
Telehealth-delivered enhanced CBTi (integrated with a sleep diary app, a therapist dashboard, and data from IoT devices) will be compared to standard telehealth CBTi and to usual treatment with sleep hygiene education. The investigators will determine effects on insomnia (primary outcome) and on clinical sleep metrics (secondary outcome), among other outcomes including cognitive performance, blood biomarkers of ADRD, and therapeutic adherence.

After screening consent and qualification, informed consent, and adherence evaluation with ambulatory devices (1wk), study participants are pseudo-randomized into one of 3 study arms (2:2:1, Enhanced CBTi : Standard CBTi : Sleep Hygiene). The living space of participants is equipped with IoT data collection devices. Participants take surveys related to sleep, have blood drawn, wear ambulatory devices, complete cognitive evaluations, and interact with nearable living space devices and an iPhone interface during a preparation week leading up to an intake telehealth appointment. Baseline data collection (1wk) occurs. Participants then adhere to behavioral therapy directives prescribed at weekly telehealth sessions with a clinically qualified therapist, take surveys related to sleep, complete cognitive evaluations, wear ambulatory devices, and interact with nearable living space devices and an iPhone interface throughout the study intervention period of 6 weeks. During the final week (coinciding with the 6th intervention week), participants have a second blood draw and return all study equipment/devices at the conclusion of participation.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speaker/reader
* Resident of the state/commonwealth of Pennsylvania for tax purposes
* Ability to complete (sign) own consent form
* Age 60-90 (inclusive, at enrollment)
* Independent Living status (or equivalent; if dwelling in a community living facility)
* Insomnia Severity Index (ISI) screening survey score of >=11
* Willing to refrain from initiating new therapeutic insomnia interventions that are not a part of this study protocol for the duration of study participation
* Willing to maintain existing physician-directed intervention for issues pertaining to sleep for the duration of study participation
* Has a residence with access to WiFi

Exclusion Criteria:

* Has a pacemaker
* Illicit drug use in the past month
* Diagnosed serious mental health disorder (e.g. psychosis or bipolar depression)
* Currently engaged in evidence-based psychotherapy for Insomnia (e.g. CBTi)
* Cohabiting with a current or previous participant in this study
* Evidence of Cognitive Impairment (a score of <18 on the abbreviated Montreal Cognitive Assessment [MoCA] screening evaluation)

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | Screening (at enrollment qualification) and Weekly (each of study weeks 1-8)
  Subjective patient completion of the Insomnia Severity Index survey. Sum of survey item responses; Minimum score: 0; Maximum score: 28. Higher sum score indicates a greater number of, or more severe, insomnia symptoms; reduction in sum score suggests improvement of insomnia.

SECONDARY OUTCOMES:
Change in Sleep Maintenance Efficiency | Nightly (each night throughout study weeks 1-8)
  Objective ambulatory activity (actigraphy) and other biometric data will be collectively used to determine sleep state. From sleep state data, Sleep Maintenance Efficiency will be calculated (i.e. percentage of time between sleep onset and awakening for the main sleep period that is spent in the sleep state). Minimum score: 0% (i.e. no sleep); Maximum score: 100% (i.e. no awake time during the sleep window). Higher percentage score indicates that a greater proportion of the rest interval was spent actually asleep; increase in percentage score suggests improvement in sleep quality.
Change in Total Sleep Time | Nightly (each night throughout study weeks 1-8)
  Objective ambulatory activity (actigraphy) and other biometric data will be collectively used to determine sleep state. From sleep state data, Total Sleep Time will be calculated (i.e. total minutes of nocturnal sleep). An increase in sleep time indicates improvement in sleep quantity.
Change in Self-Reported Sleep | Daily (each morning throughout study weeks 1-8)
  Subjective sleep diary data will be used to determine perceived sleep features (duration, quality, etc).

OTHER OUTCOMES:
Change in cognitive test battery performance | Daily: Baseline (throughout 1st-2nd study weeks) and Post-Treatment (throughout 8th study week)
  Objective test performance metrics on an ambulatory cognitive test battery delivered with a smartphone device.
Adherence to clinical therapeutic prescription | Daily: during Intervention (throughout 3rd-7th study weeks) and Post-Treatment (throughout 8th study week)
  Attendance and completion of clinically assigned behavioral tasks (subjective patient self-report and evidence from objective data from ambulatory and nearable IoT devices).
Change (pg/mL) in blood biomarkers of Alzheimer's-related dementia and Inflammation | Baseline (week 2) vs. Post-Treatment (8th week)
  Blood biomarkers suggestive of Alzheimer's disease and related dementias (ADRD), including beta-amyloid (Aβ), Tau, Neurofilament Light chain protein, glial fibrillary acidic protein (GFAP), and brain-derived neurotrophic factor (BDNF). Blood biomarkers indicative of inflammation, including tumor necrosis factor-alpha (TNFα) and Interleukin inflammatory cytokines.
Change in C-reactive Protein (CRP; mg/L) | Baseline (week 2) vs. Post-Treatment (8th week)
  C-reactive Protein (CRP), a blood biomarker indicative of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Taylor, Ph.D., Principal Investigator — The University of Arizona; Daniel Gartenberg, Ph.D., Principal Investigator — Sleep Space, Inc.; Orfeu M Buxton, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No